CLINICAL TRIAL: NCT07299903
Title: The Effect of Information, Motivation, Behavioral Skills (IMB) Model-Based Sleep Hygiene Education on Sleep Quality and Depression Level in Menopausal Women: A Methodological and Experimental Study
Brief Title: IMB-Based Sleep Hygiene Education for Menopausal Women: Effects on Sleep Quality and Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20.11.2025-09/1541
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Insomnia; Depressive Symptoms
Keywords: Menopause; Sleep quality; Sleep hygiene; Depression; Women's health; Randomized controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Sleep Hygiene

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Hygiene Education (Experimental): Participants will receive sleep hygiene education based on the Information-Motivation-Behavioral Skills (IMB) Model. Sleep habits, routines, and behaviors to improve sleep quality will be taught. Sleep quality and depression will be measured before and after the intervention, and participants will maintain daily sleep logs.
  Interventions: Behavioral: Sleep Hygiene Education
- Control (No Intervention): Participants will receive standard care without additional sleep hygiene education. Sleep quality and depression will be measured at the same time points as the intervention group.

INTERVENTIONS:
Behavioral: Sleep Hygiene Education — Education based on the IMB Model targeting sleep habits, routines, and sleep hygiene behaviors to improve sleep quality.
  Arms: Sleep Hygiene Education

SUMMARY:
This study aims to evaluate the effects of sleep hygiene education on sleep quality and depression in women during menopause. Women will be randomly assigned to either an education group or a control group. The education group will receive training based on the Information-Motivation-Behavioral Skills (IMB) Model. Sleep quality and depression levels will be measured before and after the education. The results will provide insight into whether sleep hygiene education can improve sleep quality and reduce depression in menopausal women.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of sleep hygiene education on sleep quality and depression in menopausal women. The study will be conducted in two phases. In the first phase, a menopause-specific sleep quality scale will be developed to assess sleep habits, nighttime awakenings, sleep disruptors, and sleep hygiene behaviors in this population. In the second phase, participants will be randomly assigned to either a control group or an intervention group receiving sleep hygiene education based on the Information-Motivation-Behavioral Skills (IMB) Model. Sleep quality and depression levels will be measured before and after the intervention using validated psychological and physiological assessments. Daily sleep tracking logs will also be used to monitor adherence and intervention effectiveness. The findings will provide insight into whether sleep hygiene education can improve sleep quality and reduce depression among menopausal women, and will serve as a resource for developing nursing interventions and informing health policies.

ELIGIBILITY:
Inclusion Criteria:

* Being in menopause
* Being between 40 and 60 years of age
* Having a low sleep quality score according to the Menopause-Specific Sleep Quality Scale.
* Being willing to participate in the study.
* Having no physical or mental disabilities that would hinder communication.
* Having technology (smartphone, tablet, or computer) with internet access and the ability to participate in online training.

Exclusion Criteria:

* Having a history of receiving psychological support.
* Having been diagnosed with a chronic psychiatric illness (previously diagnosed depression, anxiety disorder, etc.).
* Having a neurological or chronic systemic illness that may affect sleep quality.
* Being treated for a sleep disorder (receiving medication or psychotherapy).
* Receiving hormone replacement therapy (HT).
* Having received sleep hygiene training/therapy within the last 6 months.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | Baseline and 10 weeks after intervention
  Change in sleep quality measured using the Menopause-Specific Sleep Quality Scale before and after the sleep hygiene education intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Ayten ARIÖZ DÜZGÜN, Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
IPD Sharing Plan: Yes. De-identified IPD (protocol, SAP, and raw outcome datasets for MSSQS and BDI) will be shared with researchers submitting a methodologically sound proposal. Data will be available starting 9 months post-publication and for 36 months. Access requires a signed Data Access Agreement (DAA). Contact the Principal Investigator at [busrakaragol22@gmail.com] for proposals.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Start Date9 months following article publication End Date36 months following article publication
Access Criteria: Access is limited to qualified external researchers who submit a methodologically sound research proposal to the Principal Investigator at [busrakaragol22@gmail.com].
  Researchers will access de-identified IPD (including MSSQS/BDI data, Protocol, SAP, and Analytic Code).
  Access is conditional upon two requirements:
  Execution of a Data Access Agreement (DAA).
  Provision of ethical approval (IRB/IEC) for secondary analysis from the requester's institution.
  Data is strictly for non-commercial use.